CLINICAL TRIAL: NCT00452803
Title: A Randomized Phase II Study Preoperative Chemotherapy Versus Preoperative Concurrent Chemoradiotherapy for Patients With Biopsy-Proven N2 Stage IIIA Non-Small Cell Lung Cancer
Brief Title: Pre-operative Chemotherapy Versus Concurrent Chemoradiotherapy in N2 Positive IIIA Non Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Heung Tae Kim, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-06-164
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-07

CONDITIONS: Lung Cancer
Keywords: Non small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- study arm (Active Comparator): pre-operative chemotherapy (Pac/Cis)
  Interventions: Drug: chemotherapy
- study arm 2 (Active Comparator): Pre-operative concurrent chemoradiation therapy
  Interventions: Drug: Concurrent chemoradiation therapy; Radiation: Concurrent chemoradiation therapy

INTERVENTIONS:
Drug: chemotherapy — Paclitaxel 90mg/m2 + Cisplatin 40mg/m2 on D1 & 8 q 3weeks, Pre-OP & post-op : 2cycles (total 4 cycles)
  Arms: study arm
Drug: Concurrent chemoradiation therapy — Paclitaxel 50mg/m2 + Cisplatin 20mg/m2 on D1 & 8 q 3weeks, Pre-OP & post-op : 2cycles (total 4 cycles)
  Arms: study arm 2
Radiation: Concurrent chemoradiation therapy — Preoperative Thoracic radiation: 180cGy/fx, total: 4500cGy, 25fx
  Arms: study arm 2

SUMMARY:
It is suggested that a bimodal or trimodal approach combining neoadjuvant chemotherapy with or without radiotherapy followed by surgery provides a potentially superior method of enhancing resectability and improving locoregional control and survival compared to radiotherapy alone followed by surgery. Unsolved questions are the identification of the best induction strategy, the impact of surgery on long-term survival, and the contribution of radiation therapy in this setting. Thus, the investigators conduct a phase II trial to compare neoadjuvant chemotherapy with concurrent chemoradiotherapy in patients with biopsy proven N2 stage IIIA NSCLC to address optimal induction strategy.

DETAILED DESCRIPTION:
Preoperative Therapy Arm 1. (preoperative chemotherapy) Paclitaxel (90 mg/m2)on day 1 and 8 Cisplatin (40 mg/m2)on day 1 and 8. q 3 weeks, 2 cycles

Arm 2. (preoperative chemoradiotherapy) Paclitaxel (50 mg/m2)on day 1, 8, 15, 22 & 29 Cisplatin (20 mg/m2)on day 1, 8, 15, 22 & 29. Thoracic radiation therapy (TRT) 1.8 Gy daily, five times per week (45 Gy target dose in 5 weeks).

Postoperative Consolidation Chemotherapy:

Paclitaxel (90 mg/m2) on day 1 and 8. Cisplatin (40 mg/m2) on day 1 and 8. q 3weeks, 2 cycles

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic diagnosis of non-small cell lung cancer.
2. Presence of biopsy-proven N2 stage IIIA, according to the American Joint Committee on Cancer (AJCC), with none of the mediastinal lymph nodes > 3 cm in largest diameter.
3. Tumor amenable to surgical resection.
4. At least one unidimensional measurable lesion meeting Response Evaluation Criteria in Solid Tumors (RECIST. 2000).
5. No prior tumor therapy (surgery, radiotherapy, chemotherapy, immunotherapy, or any other type of tumor therapy).
6. Performance status of 0-1 on ECOG scale.
7. At least 18 years old.
8. Patient compliance that allows adequate follow-up.
9. Medical fitness of patients adequate for radical NSCLC surgery.
10. Adequate organ function including the following:Adequate hematologic function: WBC count ≥ 4,000/uL, absolute neutrophil count (ANC) ≥ 1,500/uL, platelet count ≥ 100,000/uL, and hemoglobin ≥ 10 gm/dL.Adequate hepatic function: bilirubin ≤ 1.5 x UNL, ALT or AST ≤ 2.5 x UNL.Adequate renal function: creatinine ≤ 1.5mg/dL.
11. Signed informed consent from patient or legal representative.12. Patients with reproductive potential must use an approved contraceptive method during and for 3 months after the study. Females with childbearing potential must have a negative urine hCG test within 7 days prior to study enrollment.

Exclusion Criteria:

1. Concurrent administration of any other tumor therapy, including radiotherapy, chemotherapy, immunotherapy.
2. Active uncontrolled infection.
3. Serious concomitant disorders that would compromise the safety of patient or compromise the patient's ability to tolerate therapy.
4. MI within preceding 6 months or symptomatic heart disease including unstable angina, congestive heart failure, or uncontrolled arrhythmia.
5. Significant neurological or mental disorder.
6. Second primary malignancy.
7. Pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2006-04; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To estimate the time to recurrence | The interval from the date of randomization to the date to the date of the first objective evidence of recurrence or to the date of death, if before recurrence

SECONDARY OUTCOMES:
To estimate the overall survival | from the date of randomization to the date of death
To assess the pathologic complete response rate and the complete resection rate | After surgery
To estimate toxicities | from the first date of treatment to 30 days after the last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Heung Tae Kim, M.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea